CLINICAL TRIAL: NCT03771183
Title: National Retrospective Study to Characterize LOng REsponder Under EribuLINE (HALAVEN®) Metastatic Breast Cancer Patients
Brief Title: Loreline Study: Characterization of Long Responders Under Eribuline
Acronym: Loreline
Status: Completed | Type: Observational
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A03054-51
Record Dates: First submitted 2018-11-28; First posted 2018-12-11 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer Patients; Therapy Related Tumor
MeSH Terms: conditions — Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients in long response during Halaven® treatment — Data collection

SUMMARY:
There is currently no strict recommendations for the management of patients who have received at least one or two lines of anthracyclines-based chemotherapy and taxane therapy for advanced breast cancer. However, Halaven® can represent a therapeutic alternative at this stage of the disease.

Indeed, since march 2011, Halaven® has been granted Marketing Authorization (MA) for patients with metastatic or locally advanced breast cancer, whose disease has progressed after at least two lines of chemotherapy for advanced disease (3rd line). In these patients, the indication for marketing authorization specifies that the previous treatment must have included an anthracycline and a taxane except in patients who can not receive these treatments.

An extension of indication was obtained on 27/06/2014 with a marketing authorization obtained in the treatment of locally advanced or second-line metastatic breast cancer.

According to the Transparency Commission of the High Authority of Health (HAS dated September 23, 2015), Halaven® (Eribulin), administered as monotherapy, in the third line of treatment and beyond, represents a therapeutic option, because it brings an improvement of medical service rendered compared to Capecitabine (XELODA®) and Vinorelbine (NAVELBINE®).

In addition, Halaven® (Eribuline) administrated as monotherapy in second-line of treatment is an alternative to other monotherapies recommended for the treatment of locally advanced or metastatic relapsed breast cancer, such as Capecitabine (XELODA®). and Vinorelbine (NAVELBINE®). But, no improvement of medical service rendered has been reported in second line of treatment.

According to these results, it would be interesting to have additional data concerning the use of Halaven® (Eribulin), in the second and third lines, but also in the fourth line.

For this purpose, the investigators propose to perform a study in patients with metastatic breast cancer who have failed treatment after the first line and beyond.

In this study, the investigators will be particularly interested in "long-responder" patients, that is to say, in objective response or with stability for 6 months or more under Halaven®, in order to better characterize these patients. Patients must have been treated by Halaven between September 2011 and December 2016, to have a sufficient follow-up for the survival data of the patients.

DETAILED DESCRIPTION:
The investigators will perform a cross-sectional study in patients with metastatic breast cancer who have failed treatment after the first line and beyond.

In this study, the investigators will be particularly interested in "long-responder" patients, that is to say, in objective response or with stability for 6 months or more under Halaven®, in order to better characterize these patients. Patients must have been treated by Halaven between September 2011 (the year of obtaining the MA in the 3rd line of treatment) and December 2016, to have a sufficient follow-up for the survival data of the patients.

The investigators will also focus on patients with liver metastases because there is limited data in this population.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 75 years
* Metastatic breast cancer patient
* Patients treated by Halaven® in second, third or fourth line of treatment for their metastatic breast cancer
* Halaven® treatment must have been received between September 2011 and December 2016
* Patients responding or in stability during at least 6 months under Halaven® treatment
* Patients pretreated by at least one line of any other chemotherapy
* Non opposition form dated and signed by the investigator (attesting that the patient consented orally that clinical, biological and imaging data concerning her were analyzed in this study)

Exclusion Criteria:

* Male
* Patient with cognitive and psychiatric disorders
* Patient deprived of liberty by judicial or administrative decision
* Insufficient knowledge or understanding of the French language which does not allow for the non-opposition form to be understood

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients will be included in order to have an homogeneous group
Study Population: This is a nationale, multicentric, retrospective study in which will be inclused metastatic breast cancer patients treated by Halaven® in second, third line or fourth line.
  Only "long responder" patients treated by Halaven®, since Septembre 2011 to December 2016, will be included in this study.
  A patient will be considered as " long responder " if she is in objective response or stability for 6 months or more from the start of Halaven® treatment
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Measure patient's age at the beginning of Halaven® treatment in patients who received Halaven® and who were in response since 6 months or more | up to at least 6 months after Halaven® start
  -patient's age at the beginning of Halaven® treatment
Characterize tumor of patients who received Halaven® and who were in response since 6 months or more | up to at least 6 months after Halaven® start
  histological tumoral type
Characterize patients who received Halaven® and who were in response since 6 months or more, according to previous treatments (neoadjuvant and/or adjuvant treatments) | up to at least 6 months after Halaven® start
  number of patients who have received neoadjuvant treatments number of patients who have received adjuvant treatments
Characterize patients who received Halaven® and who were in response since 6 months or more, according to the number of lines of treatment received for metastatic disease | up to at least 6 months after Halaven® start
  -number of lines of treatment received for metastatic disease, including treatment received before Halaven®
Characterize metastatic localizations of patients who received Halaven® and who were in response since 6 months or more | up to at least 6 months after Halaven® start
  number of patients with metastatic localizations
Characterize patients who received Halaven® and who were in response since 6 months or more | up to at least 6 months after Halaven® start
  number of patients with liver metastasis, surgery of liver metastasis
Measure the number of Halaven® injections to obtaine the "best" response in patients who received Halaven® and who were in response since 6 months or more | up to at least 6 months after Halaven® start
  -number of Halaven® injections until the " best " response is obtained
Measure the best response under Halaven® in patients who received Halaven® and who were in response since 6 months or more | up to at least 6 months after Halaven® start
  -duration of the " best " response under Halaven® (in months)
Measure hormonal receptors tumours of patients who received Halaven® and who were in response since 6 months or more | up to at least 6 months after Halaven® start
  hormonal receptors of primitive tumor (percentage of stained cells)
Measure KI-67 tumours of patients who received Halaven® and who were in response since 6 months or more | up to at least 6 months after Halaven® start
  -pathology of primitive cancer : ki-67
Measure Scarff Bloom Richardson grade tumours of patients who received Halaven® and who were in response since 6 months or more | up to at least 6 months after Halaven® start
  -pathology of primitive cancer : Scarff Bloom Richardson grade The Scarff Bloom Richardson garde will be measured with a scale from I to III. A grade III represent a worse outcome.

SECONDARY OUTCOMES:
Measure Percentage of long responders patients under Halaven® among patients treated by Halaven® in second, third and fourth line of treatment | up to at least 6 months after Halaven® start
  Percentage of patients in objective response or in stability during 6 months and more since the beginning of Halaven® treatment among all patients treated by Halaven® (in second, third and fourth line of treatment). This percentage will be collected in each participating center at the end of the study.
-Evaluate the percentage of patients with hepatic metastases | up to at least 6 months after Halaven® start
  -Percentage of liver metastatic patients
-Evaluate the specific response and/or stability in patients with hepatic metastases, that is measure percentage of liver metastatic patients in complete or partial response or in stability under Halaven® | up to at least 6 months after Halaven® start
  -Percentage of liver metastatic patients in complete or partial response or in stability under Halaven®
-Evaluate toxicities due to the use of Halaven® | up to at least 6 months after Halaven® start
  Number and percentage of patients who have a grade 3 and a grade 4 toxicity (for each toxicity reported)
  -Collection of toxicities under Halaven® Toxicities considered are toxicities grade 3, 4 and 5 (CTCAE V4.03 dated on june 14, 2010) : nausea, vomiting,diarrhea, neutropenia, anemia, leucopenia, fatigue, peripheral neuropathy, alopecia, loss of apetite. If others toxicities appear, they will be notified in the e-CRF.
-Evaluation of percentage of patients in complete or partial response or in stability under Halaven® according to number of previous metastatic treatment lines | up to at least 6 months after Halaven® start
  -Percentage of patients in complete or partial reponse or in stability under Halaven®. This percentage will be calculated in patients treated by Halaven® in second, third or fourth line of treatment
-Evaluation of Progression Free Survival (PFS) | up to at least 6 months after Halaven® start
  -Measure of time to progression (in months or in years) The PFS will be calculated from date of Halaven start to first progression date whatever the type of progression (local progression, progression of a previous metastasis and/or appearance of new metastasis, and/or new cancer).
Evaluation of overall survival | up to at least 6 months after Halaven® start
  Measure of overall survival (in months or in years) Overall survival calculated from start of Halaven to death, whatever the cause, or date of last consultation if patients are alive at the 12/31/2017.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Ange MOURET-REYNIER, MD, Principal Investigator — Centre Jean Perrin
Locations (5):
- France (5):
  - CHRU Jean Minoz, Besançon
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No